CLINICAL TRIAL: NCT04528589
Title: To Repeat or Not Repeat - A Mixed Methods Pilot Study of Patients' and Therapists' Experience With Prenatal Psychotherapy to Prevent Intergenerational Transfer of Adverse Childhood Experiences
Brief Title: To Repeat or Not to Repeat - Preventing Intergenerational Transfer of Adverse Childhood Experiences
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Marianne Aalberg, Researcher, University Hospital, Akershus
Other Study IDs: 97191
Record Dates: First submitted 2020-07-16; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Psychological Trauma
Keywords: Mother-child relations; parenting; reflective function; child development; psychotherapy
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers: Women with adverse childhood experiences referred for treatment in gestational week 20-30
  Interventions: Other: prenatal psychotherapy
- Therapists: Clinicians with experience of providing psychotherapy to women with adverse childhood experiences referred for treatment during pregnancy

INTERVENTIONS:
Other: prenatal psychotherapy — Prenatal psychotherapy to break intergenerational risk of adverse childhood events
  Groups: Mothers

SUMMARY:
The main aim of the study is to examine patients' and therapists' experiences with prenatal psychotherapy provided to pregnant women with adverse childhood experiences and how this may influence intergenerational transmission of risk. The investigators will explore a) participants' perspectives on what promoted or prevented change in psychotherapy, b) how the mothers' reflective function changes and possible factors associated with change in reflective function. Up to 20 clinically referred women in gestational week 20-30 will be included and assessed with qualitative interviews and questionnaires at the beginning of treatment and when the baby is 4 months old. The quality of the mother-infant relationship will be assessed. Seven therapists will be interviewed with a qualitative interview schedule. Outcomes of the study will inform individual tailoring of psychotherapy for a high risk group of patients and provide increased knowledge about how intergenerational risk factors change during treatment.

DETAILED DESCRIPTION:
Even with the best evidence-based treatments, one is often unsuccessful in stopping intergenerational transfer of trauma, abuse, and neglect. The implications for the next generation are severe, affecting physical and emotional health, cognitive development, and relational functioning. The perinatal phase may provide a window of opportunity in efforts to prevent intergenerational transfer of risk factors associated with adverse childhood events. There is a great need for more knowledge about how generational patterns develop and are affected by psychotherapy during pregnancy, infancy and early childhood. Little is known about patients' experiences with prenatal psychotherapy and such knowledge can inform better tailoring of treatment. The present study is the first step of a planned longitudinal study to explore the role of mothers' adverse childhood experiences and child development.

The primary aim of the study is to explore patients' experiences with prenatal psychotherapy provided to pregnant women with adverse childhood experiences and their perspectives of what promotes or hinders change in treatment. Second, aims of the study are to explore a) therapists' experiences with psychotherapy for mothers with adverse childhood experiences, and b) explore the development of intergenerational risk factors. Additionally the investigators will explore the mothers' reflective function during the course of treatment, the role of adverse and benevolent childhood memories, and mother-infant interaction when the infant is four months old. Reflective function seems to be a key factor associated with quality of care in spite of adverse events. Understanding factors associated with possible change in reflective function is thus highly important. Up to 20 clinically referred women in gestational week 20-30 will be recruited. Participants will be assessed at the beginning of therapy and when the child is four months old. A combination of quantitative measures and qualitative interviews will be used. The infant will be assessed with the neonatal assessement scale at age 4-8 weeks and the quality of the mother-infant relationship will be assessed using Parent-Child Relation Assessment at four months. In addition, seven therapists will be interviewed about their experiences providing psychotherapy for this group of high risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically referred women in gestational week 20-30
* Adverse Childhood Experiences Questionnaire (ACE) score of 2 or more

Exclusion Criteria:

* Known IQ below 70
* Ongoing substance abuse
* Planned referral to mother-child center after birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Study Population: Mothers: Clinically referred pregnant women with adverse childhood experiences. Therapists: Therapists providing prenatal psychotherapy to women with adverse childhood experiences
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Experiences with prenatal psychotherapy | 4 months after birth
  Qualitative interview conducted 4 months after birth examining the mothers' experiences with the treatment

SECONDARY OUTCOMES:
Maternal Reflective functioning - Parent Development Interview | Gestational week 20-30 to 4 months after birth
  Assessment of change in mother's reflective functioning
Therapists' experiences with providing psychotherapy for women with adverse childhood events | Through study completion, an average of 1 year
  A qualitative interview examining positive and negative experiences with providing prenatal psychotherapy to women to prevent intergenerational transmission of adverse childhood events

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Aalberg, Phd, Principal Investigator — University Hospital, Akershus
Locations (1):
- BUP Øvre Romerike, Jessheim, Norway

IPD SHARING:
Plan to Share IPD: No